CLINICAL TRIAL: NCT07126288
Title: A Phase II/III, Seamless, Multicenter, Randomized, Open-Label, Positive-Comparator Controlled Clinical Trial to Evaluate the Efficacy and Safety of GB08 Injection in Pediatric Patients With Growth Hormone Deficiency
Brief Title: Evaluating the Efficacy and Safety of GB08 Injection in Pediatric Patients With Growth Hormone Deficiency
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shenzhen Kexing Pharmaceutical Co., Ltd. (Network)
Responsible Party: Sponsor
Organization: Kexing Biopharm Co., Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: KXZY-GB08-201
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Growth Hormone Deficiency in Children; Growth Hormone Deficiency (GHD); Growth Hormone
Keywords: growth hormone deficiency; annualized height velocity; growth hormone; clinical trial; GB08 injection
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone

STUDY DESIGN:
Intervention Model Description: Phase II/III seamless design clinical study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PhaseII GB08 0.4 mg/kg (Experimental): GB08 0.4mg/kg subcutaneous injection, once a week for 24 weeks
  Interventions: Drug: GB08
- PhaseII GB08 0.8 mg/kg (Experimental): GB08 0.8mg/kg subcutaneous injection, once a week for 24 weeks
  Interventions: Drug: GB08
- PhaseII GB08 1.2 mg/kg (Experimental): GB08 1.2mg/kg subcutaneous injection, once a week for 24 weeks
  Interventions: Drug: GB08
- PhaseII Norditropin NordiFlex (Active Comparator): Norditropin NordiFlex 0.035 mg/kg subcutaneous injection, daily, for 24 weeks
  Interventions: Drug: Norditropin NordiFlex
- PhaseIII GB08 (Experimental): GB08 subcutaneous injection (The dose will be determined by data from PhaseII), once a week for 52 weeks
  Interventions: Drug: GB08
- PhaseIII Norditropin NordiFlex (Active Comparator): Norditropin NordiFlex 0.035 mg/kg subcutaneous injection, daily, for 52 weeks
  Interventions: Drug: Norditropin NordiFlex

INTERVENTIONS:
Drug: GB08 — In Phase II trial, eligible PGHD patients will receive GB08 0.4mg/kg, 0.8mg/kg, or 1.2mg/kg subcutaneous injection, once a week for 24 weeks.
  In Phase III trial, the individuals will receive GB08 subcutaneous injection, once a week for 52 weeks. The dose of GB08 at this stage will be determined by the outcomes of Phase II.
  Arms: PhaseII GB08 0.4 mg/kg; PhaseII GB08 0.8 mg/kg; PhaseII GB08 1.2 mg/kg; PhaseIII GB08
Drug: Norditropin NordiFlex — Norditropin NordiFlex 0.035 mg/kg subcutaneous injection, daily, for 24 weeks (Phase II) or 52 weeks (Phase III)
  Arms: PhaseII Norditropin NordiFlex; PhaseIII Norditropin NordiFlex

SUMMARY:
This study aims to evaluate the efficacy and safety of GB08 injection compared to Norditropin NordiFlex in pediatric patients with growth hormone deficiency (PGHD). It seeks to resolve the following questions:

* 1: Does GB08 injection demonstrate comparable efficacy in treating PGHD at 24 weeks compared to Norditropin NordiFlex?
* 2: Which dose (0.4 mg/kg, 0.8 mg/kg, and 1.2 mg/kg) of GB08 injection best balances efficacy and safety in treating PGHD at 24 weeks?
* 3: Does GB08 injection maintain its efficacy in treating PGHD at 52 weeks compared to Norditropin NordiFlex? To achieve these, GB08 injection will be compared to Norditropin NordiFlex to see if it provides a more effective or safer treatment option for PGHD.

This is a Phase II/III, Seamless, Multicenter, Randomized, Open-Label, Positive-Comparator Controlled Clinical Trial with two stages. Stage 1 answers questions #1 and #2 by comparing the efficacy and safety of GB08 injection and Norditropin NordiFlex intervention among PGHD at 24 weeks. It involves four groups (n=16 each): GB08 0.4 mg/kg, GB08 0.8 mg/kg, GB08 1.2 mg/kg, and Norditropin NordiFlex 0.035 mg/kg. GB08 and Norditropin NordiFlex will be administered once weekly and once daily, respectively. The primary outcome measurement is annualized height velocity (AHV) at 24 weeks. Other measurements include growth hormone levels, safety parameters, immunogenicity markers, and pharmacokinetic/pharmacodynamic profiles.

The optimal GB08 dose will be further investigated in Stage 2, which answers question #3. At this stage, PGHD patients will randomly receive either GB08 injection or Norditropin NordiFlex intervention for 52 weeks (n=102 for each). After that, the efficacy and safety of GB08 will also be detected.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, positive-controlled Phase II/III seamless design clinical study evaluating the efficacy and safety of GB08 injection in pediatric patients with growth hormone deficiency (PGHD). It aims to compare the efficacy and safety of GB08 injection with Norditropin NordiFlex in PGHD patients, thereby benefiting this population. This study involves two parts: Phase II and Phase III.

Phase II: Identifying the Optimal Dose This part assesses the efficacy and safety of three doses of GB08 in treating PGHD to recommend the optimal dose for the phase III.

Eligible patients with PGHD will be randomly divided into four groups (n=16 per group) and stratified by GH peak value (≤5 μg/L and >5 μg/L). They will receive GB08 0.4 mg/kg, GB08 0.8 mg/kg, GB08 1.2 mg/kg, or Norditropin NordiFlex 0.035 mg/kg (positive control) treatment for 24 weeks with another 28 weeks of follow-up. GB08 and Norditropin NordiFlex therapy will be provided once weekly and once daily, respectively. All participants will have blood samples collected for pharmacokinetics (GB08 groups only), pharmacodynamics, immunogenicity, and safety and efficacy assessments, as well as records of concomitant medications/treatments and adverse events. The primary outcome measurement is the annualized height velocity (AHV) at 24 weeks among the four groups. The optimal GB08 dose will be identified based on the 24-week data.

Phase III: The 52-week efficacy and safety of GB08 injection compared to Norditropin NordiFlex This part aims to evaluate the efficacy of GB08 injection compared to Norditropin NordiFlex in PGHD patients at 52 weeks.

It contains a treatment group (GB08 injection) and a control group (Norditropin NordiFlex), each with 102 participants. Accordingly, they will receive GB08 or Norditropin NordiFlex intervention for 52 weeks. The dose of GB08 will be determined by Phase II. Stratified randomization will be based on age (<6 years vs. ≥6 years), gender (male vs. female), and GH peak value (≤ 5 ug/L, 5-7 ug/L, >7 ug/L). The treatment period will last for 52 weeks with a 2-week follow-up. The primary endpoint measurement is the efficacy of GB08 injection at the 52nd week compared to Norditropin NordiFlex.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Growth Hormone Deficiency (GHD) based on medical history, clinical symptoms and signs, GH stimulation tests, and imaging studies. The participant must meet the following:

1. Absolute height 2 standard deviations (SD) below the mean height of children of the same age and sex, according to the standardized growth curves for children and adolescents in China (0-18 years old) published in 2009.
2. Annualized height velocity (AHV) ≤ 5.0 cm/year, calculated from measurement of 6 to 18 months before screening.
3. GH peak ≤ 10 ng/ml proved by two different GH stimulation tests within a year before screening.
4. Bone age lagging at least 1 year behind actual age (bone age assessment within the past 6 months before screening), with girls < 10 years old and boys < 11 years old.

2. Aging > 3 years and ≤ 10 years (girls) or ≤ 11 years (boys) based on birth date; Tanner stage I (testicular volume < 4 ml for boys and no palpable breast tissue for girls) 3. Uniform short stature with normal intellectual development. 4. IGF-1 levels below the mean for children and adolescents of the same age and sex, at least 1 SD below (IGF-1 SDS ≤ -1.0).

5. Body mass index (BMI) within ±2 SD of the mean BMI for children and adolescents of the same age and sex.

6. For subjects with GHD as part of multiple pituitary hormone deficiencies, must be stable for ≥1 month, as determined by the investigator.

7. Guardians understand and sign the Informed Consent Form (ICF). If the participant is ≥8 years old, they must also sign the ICF. For participants <8 years old who can express consent, their consent must be recorded.

Exclusion Criteria:

1. History of systematic growth-promoting therapy, including growth hormone and sex hormones.
2. Severe allergic constitution or known allergy to growth hormone or its excipients, such as mannitol, lysine, or sodium chloride.
3. Closed epiphyses.
4. Other types of growth disorders such as idiopathic short stature, Turner syndrome, Noonan syndrome, Prader-Willi syndrome, and Russell-Silver syndrome.
5. Short stature due to other causes, such as intrauterine growth restriction, familial short stature, thyroid hormone deficiency, adrenal insufficiency, antidiuretic hormone deficiency, celiac disease, rickets, psychological factors, chronic kidney disease, infections, or trauma.
6. Any clinically significant abnormalities that may affect growth or growth assessment; subjects with liver or kidney dysfunction (ALT > 1.5 times upper limit of normal, creatinine > upper limit of normal), chronic diseases (malnutrition, fasting blood glucose ≥ 126 mg/dL or HbA1c ≥ 6.5%), diabetes, severe cardiac, pulmonary, hematological, or systemic infections, immunodeficiency, psychiatric disorders, or congenital malformations.
7. Infectious diseases, such as hepatitis B, hepatitis C, AIDS, syphilis, or tuberculosis (HBV surface antigen-positive subjects must undergo HBV DNA testing; HCV antibody-positive subjects must undergo HCV RNA testing; if HBV DNA or HCV RNA > detection limit, they are excluded).
8. Use of corticosteroids or other steroids within the past 12 months, such as long-term steroid use for asthma.
9. History of pituitary or hypothalamic tumors, or other intracranial tumors on MRI; history of leukemia, lymphoma, or other malignancies.
10. History of radiation therapy or chemotherapy.
11. Congenital intracranial hypertension.
12. Femoral head slipped epiphysis (SCFE).
13. Spinal scoliosis > 15°.
14. Participation in any other drug clinical trial within the past 3 months (as a subject).
15. Other factors deemed unsuitable for participation in the study by the investigator.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — males: 3-11 years old; females: 3-10 years old
Enrollment: 268 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-12-23 (Estimated)

PRIMARY OUTCOMES:
PhaseII-Comparison of annualized height velocity at 24 weeks | From enrollment to end of treatment at 24 weeks
  Comparison of annualized height velocity of PGHD patients receiving 24-week GB08 and Norditropin NordiFlex treatment
PhaseIII-Comparison of annualized height velocity at week 52 | From enrollment to end of treatment at week 52
  Comparison of annualized height velocity between PGHD patients receiving GB08 and Norditropin NordiFlex at 52 weeks

SECONDARY OUTCOMES:
PhaseII-annualized height velocity at weeks 4, 12, 36, 48, 52 | From enrollment to weeks 4, 12, 36, 48, 52
PhaseII-Standard deviation (SD) scores of AHV of GB08 injection and Norditropin NordiFlex at baseline, and at weeks 4, 12, 36, 48, 52 | From enrollment to weeks 4, 12, 36, 48, 52
PhaseII-Standard deviation of actual height SDS (Ht SDS CA) of GB08 injection and Norditropin NordiFlex at weeks 4, 12, 24, 36, 48, 52 | From enrollment to weeks 4, 12, 24, 36, 48, 52
PhaseII-Standard deviation of bone age (BA) SDS (Ht SDS BA) of GB08 injection and Norditropin NordiFlex at week 24 and 52 | From enrollment to weeks 24 and 52
PhaseII-Tanner stage changes at baseline and at weeks 12, 24, 52 | From enrollment to weeks 12, 24, and 52
PhaseII-Body weight and BMI changes at baseline and at weeks 2, 4, 8, 12, 24, 52 | From enrollment to weeks 2, 4, 8, 12, 24, and 52
PhaseII-Ratio of BA to CA at baseline and at weeks 24, 52 | From enrollment to weeks 24 and 52
PhaseII-Serum IGF-1, IGF-1 SDS, and IGFBP-3 levels, and their changes from baseline at weeks 2, 4, 8, 12, 24, 36, 48, 52 | From enrollment to weeks 2, 4, 8, 12, 24, 36, 48, and 52
PhaseII-Serum IGF-1, IGF-1 SDS, and IGFBP-3 levels, and their changes from baseline at 48 hours post-dose of GB08 injection at weeks 2, 4, 8, 12, 24, 36, 48, 52 | From enrollment to weeks 2, 4, 8, 12, 24, 36, 48, and 52
PhaseIII-AHV of GB08 injection and Norditropin NordiFlex at baseline, and at weeks 4, 12, 24, 36, 48, 52 | From enrollment to weeks 4, 12, 24, 36, 48, and 52
PhaseIII-Standard deviation (SD) scores of AHV of GB08 injection and Norditropin NordiFlex at baseline, and at weeks 4, 12, 24, 36, 48, 52 | From enrollment to weeks 4, 12, 24, 36, 48, and 52
PhaseIII-Standard deviation of actual height SDS (Ht SDS CA) of GB08 injection and Norditropin NordiFlex at weeks 4, 12, 24, 36, 48, 52 | From enrollment to weeks 4, 12, 24, 36, 48, and 52
PhaseIII-Standard deviation of bone age (BA) SDS (Ht SDS BA) of GB08 injection and Norditropin NordiFlex at week 52 | From enrollment to week 52
PhaseIII-Tanner stage changes at baseline and at weeks 12, 24, 52 | From enrollment to weeks 12, 24, and 52
PhaseIII-Body weight and BMI changes at baseline and at weeks 2, 4, 8, 12, 24, 52 | From enrollment to weeks 2, 4, 8, 12, 24, and 52
PhaseIII-Serum IGF-1, IGF-1 SDS, and IGFBP-3 levels, and their changes from baseline at weeks 2, 4, 8, 12, 24, 36, 48, 52 | From enrollment to weeks 2, 4, 8, 12, 24, 36, 48, and 52
PhaseIII-Serum IGF-1, IGF-1 SDS, and IGFBP-3 levels, and their changes from baseline at 48 hours post-dose of GB08 injection at weeks 2, 4, 8, 12, 24, 36, 48, 52 | From enrollment to weeks 2, 4, 8, 12, 24, 36, 48, and 52
PhaseII-Safety Evaluation Endpoints | weeks 2, 4, 8, 12, 24, 36, 48, 52.
  Adverse events (AEs), vital signs, ECG, physical examination, abnormal clinical laboratory parameters (including but not limited to complete blood count, blood biochemistry, urinalysis, thyroid function, fasting insulin, prolactin, HbA1c, fasting serum cortisol), and injection site examination.
PhaseII-Immunogenicity Evaluation Endpoints | weeks 12, 24, 36, 52
  Blood samples will be collected at baseline and at weeks 12, 24, 36, 52 to determine the presence of anti-drug antibodies (ADA). If ADA is positive, neutralizing antibody and titer analysis will be performed. If ADA-positive subjects are needed for safety and efficacy analysis, additional ADA, neutralizing antibody, and titer testing may be conducted.
PhaseII-Pharmacokinetics Evaluation Endpoints | weeks 2, 4, 8, 12, 24, 36, 48, 52.
  PK parameters: maximum concentration (Cmax), area under the curve from time 0 to the last measurable concentration (AUC0-t), area under the curve from time 0 to infinity (AUC0-inf), time to peak concentration (Tmax), elimination rate constant (λz), elimination half-life (t1/2), apparent volume of distribution (Vd/F), apparent clearance (CL/F), AUC0-inf extrapolated percentage (AUC_%Extrap).
PhaseII-Pharmacodynamics Evaluation Endpoints | time 0 to 168 hours
  Observed maximum effect (Emax), time to reach maximum effect (TEmax), area under the effect-time curve from time 0 to the last measurable time point (AUEC0-t), area under the effect-time curve from time 0 to 24 hours (AUEC0-24h), area under the effect-time curve from time 0 to 168 hours (AUEC0-168h).
PhaseIII-Safety Evaluation Endpoints | weeks 2, 4, 8, 12, 24, 36, 48, 52
  Adverse events (AEs), vital signs, 12-lead ECG, physical examination, abnormal clinical laboratory parameters (including but not limited to complete blood count, blood biochemistry, urinalysis, thyroid function, fasting insulin, prolactin, HbA1c, fasting serum cortisol), and injection site examination.
PhaseIII-Immunogenicity Evaluation Endpoints | weeks 12, 24, 36, 52
  Blood samples will be collected at baseline and at weeks 12, 24, 36, 52 to determine the presence of anti-drug antibodies (ADA). If ADA is positive, neutralizing antibody and titer analysis will be performed. If ADA-positive subjects are needed for safety and efficacy analysis, additional ADA, neutralizing antibody, and titer testing may be conducted.
PhaseIII-Pharmacodynamics Evaluation Endpoints | weeks 12, 24, 36, 52
  GB08 injection and Norditropin NordiFlex concentrations of IGF-1 and IGFBP-3, relative changes from baseline, and percentage changes at baseline and at weeks 12, 24, 36, 52.

CONTACTS AND LOCATIONS:
Overall Officials: Junfen Fu, Principal Investigator — Children's Hospital of Zhejiang University School of Medicine; Yijia Zhang, Study Director — Shenzhen Kexing Pharmaceutical Co., Ltd.
Locations (16):
- China (16):
  - Xiamen Maternal and Child Health Hospital, Xiamen, Fujian
  - Nanyang Central Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Wuhan Children's Hospital, Wuhan, Hubei
  - Suzhou University Children's Hospital, Suzhou, Jiangsu
  - Jiangxi Children's Hospital, Nanchang, Jiangxi
  - Pingxiang Maternal and Child Health Hospital, Pingxiang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Linyi Maternal and Child Health Hospital, Linyi, Shandong
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Meishan People's Hospital, Meishan, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Women's and Children's Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christiansen JS, Backeljauw PF, Bidlingmaier M, Biller BM, Boguszewski MC, Casanueva FF, Chanson P, Chatelain P, Choong CS, Clemmons DR, Cohen LE, Cohen P, Frystyk J, Grimberg A, Hasegawa Y, Haymond MW, Ho K, Hoffman AR, Holly JM, Horikawa R, Hoybye C, Jorgensen JO, Johannsson G, Juul A, Katznelson L, Kopchick JJ, Lee KO, Lee KW, Luo X, Melmed S, Miller BS, Misra M, Popovic V, Rosenfeld RG, Ross J, Ross RJ, Saenger P, Strasburger CJ, Thorner MO, Werner H, Yuen K. Growth Hormone Research Society perspective on the development of long-acting growth hormone preparations. Eur J Endocrinol. 2016 Jun;174(6):C1-8. doi: 10.1530/EJE-16-0111. Epub 2016 Mar 23. PMID 27009113
- [Background] Rosenfeld RG, Bakker B. Compliance and persistence in pediatric and adult patients receiving growth hormone therapy. Endocr Pract. 2008 Mar;14(2):143-54. doi: 10.4158/EP.14.2.143. PMID 18308651
- [Background] Allen DB, Backeljauw P, Bidlingmaier M, Biller BM, Boguszewski M, Burman P, Butler G, Chihara K, Christiansen J, Cianfarani S, Clayton P, Clemmons D, Cohen P, Darendeliler F, Deal C, Dunger D, Erfurth EM, Fuqua JS, Grimberg A, Haymond M, Higham C, Ho K, Hoffman AR, Hokken-Koelega A, Johannsson G, Juul A, Kopchick J, Lee P, Pollak M, Radovick S, Robison L, Rosenfeld R, Ross RJ, Savendahl L, Saenger P, Sorensen HT, Stochholm K, Strasburger C, Swerdlow A, Thorner M. GH safety workshop position paper: a critical appraisal of recombinant human GH therapy in children and adults. Eur J Endocrinol. 2016 Feb;174(2):P1-9. doi: 10.1530/EJE-15-0873. Epub 2015 Nov 12. PMID 26563978
- [Background] Cook DM, Rose SR. A review of guidelines for use of growth hormone in pediatric and transition patients. Pituitary. 2012 Sep;15(3):301-10. doi: 10.1007/s11102-011-0372-6. PMID 22271255
- [Background] Yuen KCJ, Biller BMK, Radovick S, Carmichael JD, Jasim S, Pantalone KM, Hoffman AR. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY GUIDELINES FOR MANAGEMENT OF GROWTH HORMONE DEFICIENCY IN ADULTS AND PATIENTS TRANSITIONING FROM PEDIATRIC TO ADULT CARE. Endocr Pract. 2019 Nov;25(11):1191-1232. doi: 10.4158/GL-2019-0405. PMID 31760824
- [Background] Kim JH, Chae HW, Chin SO, Ku CR, Park KH, Lim DJ, Kim KJ, Lim JS, Kim G, Choi YM, Ahn SH, Jeon MJ, Hwangbo Y, Lee JH, Kim BK, Choi YJ, Lee KA, Moon SS, Ahn HY, Choi HS, Hong SM, Shin DY, Seo JA, Kim SH, Oh S, Yu SH, Kim BJ, Shin CH, Kim SW, Kim CH, Lee EJ. Diagnosis and Treatment of Growth Hormone Deficiency: A Position Statement from Korean Endocrine Society and Korean Society of Pediatric Endocrinology. Endocrinol Metab (Seoul). 2020 Jun;35(2):272-287. doi: 10.3803/EnM.2020.35.2.272. Epub 2020 Jun 24. PMID 32615711
- [Background] Ranke MB, Wit JM. Growth hormone - past, present and future. Nat Rev Endocrinol. 2018 May;14(5):285-300. doi: 10.1038/nrendo.2018.22. Epub 2018 Mar 16. PMID 29546874
- [Background] Cunningham BC, Ultsch M, De Vos AM, Mulkerrin MG, Clauser KR, Wells JA. Dimerization of the extracellular domain of the human growth hormone receptor by a single hormone molecule. Science. 1991 Nov 8;254(5033):821-5. doi: 10.1126/science.1948064.
- [Background] Kopchick JJ, Parkinson C, Stevens EC, Trainer PJ. Growth hormone receptor antagonists: discovery, development, and use in patients with acromegaly. Endocr Rev. 2002 Oct;23(5):623-46. doi: 10.1210/er.2001-0022. PMID 12372843
- [Background] DOI:10.3969/j.issn.2095-1736.2020.05.103.
- [Background] de Fries Jensen L, Antavalis V, Odgaard-Jensen J, Rossi A, Pietropoli A, Hojby M. Efficacy and Safety of Somapacitan Relative to Somatrogon and Lonapegsomatropin in Pediatric Growth Hormone Deficiency: Systematic Literature Review and Network Meta-analysis. Adv Ther. 2024 Nov;41(11):4098-4124. doi: 10.1007/s12325-024-02966-y. Epub 2024 Sep 11. PMID 39261416